CLINICAL TRIAL: NCT01855152
Title: An Optimized Person Centred Intervention to Improve Quality of Life for People With Dementia Living in Care Homes. A Cluster Randomized Controlled Trial.
Brief Title: Improving Well-being and Health for People With Dementia
Acronym: WHELD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: professor Clive Ballard (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, professor Clive Ballard, Chief investigator, King's College London
Organization: King's College London (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Grant RP-PG-0608
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Dementia
Keywords: Dementia; Care Homes; Quality of life; Antipsychotic medication; Behavioural symptoms; Cost effectiveness; Implementation; Person centred care; Social interaction
MeSH Terms: conditions — Dementia; Behavioral Symptoms | interventions — Health; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Optimised WHELD intervention (Experimental): The optimised WHELD intervention combining person centred care, promoting person centred activities and interactions and provide care home staff and general practitioners with updated knowledge regarding the optimal use of psychotropic medications for persons with dementia in care homes, is more effective in improving the quality of life and mental health, than usual care for people with dementia living in nursing homes.
  Interventions: Other: Optimised WHELD intervention
- Treatment as usual (Experimental): Treatments delivered as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Optimised WHELD intervention — Experimental: Optimised WHELD intervention
  Other Names: Improving Well-being and Health for People with Dementia
  Arms: Optimised WHELD intervention
Other: Treatment as usual — Treatment delivered as usual in the care home
  Arms: Treatment as usual

SUMMARY:
800,000 people in the United Kingdom (UK)have dementia, of which 250,000 are living in care homes. These individuals have complex mental health problems, disabilities and social needs, which if unmet will continue to adversely affect each individual, as well as the main goal of enabling people to "live well with dementia", as presented in the National Dementia Strategy (NDS) (Department of Health, 2009).

This optimized intervention WHELD is based on a factorial study and qualitative evaluation designed to facilitate the design of this current study and will combine this with the most effective elements of existing approaches to develop a comprehensive but practical intervention to improve quality of life in persons with dementia living in care homes. The intervention will combine training on person centred care, promoting person centred activities and interactions and provide care home staff and general practitioners with updated knowledge regarding the optimal use of psychotropic medications for persons with dementia in care homes.

The overarching goal of this trial is to determine whether this optimised WHELD intervention is more effective in improving the quality of life and mental health, than the usual care provided people with dementia living in nursing homes. The cost effectiveness of the intervention will be assessed as well, with the aim to provide a cost effective, simple and practical intervention, improving quality of life and mental health of people with dementia in care homes; which can be rolled out nationally to all UK care homes as an National Health Service (NHS) intervention. The trial will be a randomised controlled 2-arm cluster single blind trial that will take place for 9 months across 80 care homes in UK.

DETAILED DESCRIPTION:
The main objective of this current study is to determine whether the optimised WHELD intervention, will significantly improve quality of life for people with dementia in comparison to the usual care provided in care homes.

Key secondary objectives will be to determine the specific impact of the optimised WHELD intervention on a range of outcomes including mental health and unmet needs, physical health and use of psychotropic drugs, staff attitudes and the quality of the interaction of care staff with people with dementia, person centred environment in care home settings and overall provide a cost-effective, simple and practical intervention.

We hypothesise that the intervention will significantly improve several key outcomes. Specifically we hypothesise that, compared to treatment as usual the optimised WHELD intervention will:

• Improve quality of life for people with dementia living in nursing homes

The secondary hypotheses are that the optimized WHELD intervention will:

* Reduce agitation, other behavioural and neuropsychiatric symptoms
* Reduce the use of antipsychotic and other psychotropic drugs use
* Reduce unmet needs
* Reduce mortality
* Improve mood and depression
* Improve the quality of interactions between staff and residents
* Provide person centred environment in care home settings
* Provide a cost-effective intervention

The study design is a cluster randomised controlled, 2 arms trial to be run in 80 care homes, including 960 - 1280 participants.

Each cluster in the optimised WHELD intervention arm will receive the optimised WHELD intervention for 9 months.

Evaluations will be undertaken to understand the breadth of benefits conferred by the intervention to be assessed when used in comparison with the progress of the participants residing in the care homes allocated to the TAU trial arm. Baseline and follow up data will be collected on all consented residents who meet the inclusion criteria at each participating care home.

ELIGIBILITY:
Inclusion Criteria:

Care homes, which identify themselves as catering for people with dementia within its literature, in the Oxfordshire, Buckinghamshire and London localities

Care homes which demonstrate a minimum acceptable standard of care according to Care Quality Commission (CQC)

All individuals residing in participating care homes who scores '1' or greater on the Clinical Dementia Rating Scale (CDR)

Exclusion Criteria:

Less than 60% of the residents have dementia.

Receiving special support from local authority

Care home are not adequate according to CQC checks on standards of care.

Data will not be collected from individuals for whom consent has not been obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (DEMQOL-proxy) | Change in quality of life from baseline assessment point to the 9 month intervention period in both intervention and control group
  DEMQOL-Proxy (main outcome measure) is a 31 item interviewer-administered questionnaire answered by a caregiver with the score range of 31 to 124. The The measure is also validated as a method for calculating Quality Adjusted life Year (QALY) for health economic analysis.
  DEMQOL (secondary outcome measure) assesses the health-related quality of life (HRQoL) for people with dementia. The measure consists of two questionnaires. DEMQOL, conducted with person with dementia is a 28 item interviewer-administered questionnaire with the score range of 28 to 112.

SECONDARY OUTCOMES:
Quality of life in late - stage dementia (QUALID) | Change in quality of life in late stage dementia measure from baseline to the 9 months of the intervention.
  The QUALID is a reliable valid scale, administered to caregivers, for rating quality of life in people with late-stage dementia. The scale measures 11 observable behaviours indicating activity and emotional states. Ratings are made for observations made over the preceding 7 days. Items are rated on a 5-point Likert scale with QUALID scores ranging from 12 to 45 points with lower scores reflecting a higher quality of life (QOL).
Global Deterioration Scale (GDS). | The outcome measure will be assessed prior to randomization and after 9 months of the intervention.
  The GDS is a staging scale indicating deterioration in dementia, The scale details clinical descriptions of seven major distinguishable stages, ranging from normal cognition to severe dementia. Stages 1 - 3 are the pre dementia stages. Stages 4 -7 reflect the stages of dementia. People beginning with stage 5 are no longer survive without assistance.
Cohen-Mansfield Agitation Inventory (CMAI) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention
  The CMAI is a caregivers' rating questionnaire to specify agitated behaviour (Cohen-Mansfield et al, 1989). The CMAI consists of 29 items related to agitated behaviour, each of which is rated on a 7-point scale of frequency, from 1 = never to 7 = several times an hour. The rating is based on a face-to-face interview with a caregiver.
Neuropsychiatric Inventory nursing home version (NPI-NH) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention
  The NPI is a validated structured interview assessment with the informant (care staff), that assesses behavioural disturbances in patients with dementia [25]. This 12-item version consists of 10 behavioural and two neurovegetative areas. It provides both a total score as well as scores for a number of sub-scales (e.g., delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, disinhibition, elation/euphoria, apathy/indifference, irritability/lability, aberrant motor activity, sleep, and appetite/eating disorders). The frequency, severity and caregiver distress for each domain are measured. The total possible maximum score is 144. A higher score reflects increased frequency and severity of the disturbances. This specific version is developed for use in nursing homes (NPI-NH), with adapted questions in the standardized interview and the caregiver distress assessment is adapted to occupational disruptiveness.
Cornell Scale for Depression in Dementia (CSDD) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention
  The CSDD is an assessment of signs and symptoms of major depression in patients with dementia. The CSDD uses a comprehensive interviewing approach that derives information via semi-structured interviews with the participant and the care staff. Many of the items during the patient interview can be filled after direct observation of the patient. The final ratings of the CSDD items represent the rater's clinical impression rather than the responses of the informant or the patient. Each item is rated for severity on a scale of 0-2 (0=absent, 1=mild or intermittent, 2=severe). The item scores are added. Scores above 10 indicate a probable major depression. Scores above 18 indicate a definite major depression. Scores below 6 as a rule are associated with absence of significant depressive symptoms.
The Abbey Pain Scale | The outcome measure will be assessed prior to randomization and after 9 months of the intervention.
  The abbey pain scale is an observational brief indicator of pain for people with end-stage dementia. The scale is rated on six non verbal indicators of pain where 0 is none and 3 is severe.
Camberwell Assessment of Need for the Elderly (CANE Version IV) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention
  The CANE is a comprehensive assessment assessing 24 areas of social, medical, psychological, and environmental needs. The overall rating on the CANE will be based on all the information gathered throughout the structured interview with the care staff and based on the information collected through looking at the case-note reviews and observations within the care home.
Quality of Interaction Scale (QUIS) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention
  QUIS is an observational tool which measures the quality of interactions between staff and resident and personcentered environment in care home settings.
Sheffield Care Environment Assessment Matrix (SCEAM) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention
  SCEAM is a comprehensive observational assessment of the care environment, which covers items such as privacy, choice and degree of control experienced by residents. Assessors require no particular training and can carry out the assessment mostly by walking through the home and directly observing the building and the way it is used in practice. The majority of items relate to the residents, but there is also a section relating specifically to staff and the provision made for them.
Client Service Receipt Inventory (CSRI) | The outcome measure will be assessed prior to randomization and after 9 months of the intervention.
  The CSRI is used to estimate the cost of service packages for each participant in the study. Information is collected on the current living arrangements, use of hospital, community-based and day services over a defined retrospective of 3 months in this study. The data collected through the CSRI can be used to calculate service costs and total costs of care.

CONTACTS AND LOCATIONS:
Overall Officials: Bob Woods, Professor, Study Chair — Bangor University
Locations (1):
- King's College London, London, United Kingdom